CLINICAL TRIAL: NCT04076917
Title: BIO-Precision Study
Brief Title: Assessment of the Utility of BIOMONITOR to Identify Atrial Fibrillation (AF) in Ablation Candidates Using Precise AF Detection
Acronym: BIO-Precision
Status: Terminated | Type: Observational
Why Stopped: This study was terminated by the sponsor since study timelines were extended significantly due to slow enrollment, partly influenced by the COVID-19 pandemic.
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO-Precision
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate the diagnostic utility of BIOTRONIK's subcutaneous cardiac rhythm monitor for the detection of AF prior to an ablation procedure.

DETAILED DESCRIPTION:
BIO-Precision is a post-market study investigating the utility of atrial fibrillation (AF) detection using BIOTRONIK's subcutaneous cardiac rhythm monitor, BIOMONITOR. The purpose of this study is to evaluate the diagnostic utility of BIOTRONIK's BIOMONITOR for the detection and confirmation of AF prior to an ablation procedure. Study population includes patients with paroxysmal AF being evaluated for an AF ablation. Holter monitoring for 48 hours will be performed after insertion of the BIOMONITOR but prior to AF ablation. This study will enroll up to 100 subjects, to obtain 60 usable Holter recordings, at 5 study sites within the United States (U.S.). Study subjects will be followed for three months after the completion of a 48 hr Holter monitor.

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for subcutaneous cardiac rhythm monitor insertion according to local regulations
* Patient is able to understand the nature of the study and provide written informed consent
* Inserted within the prior 30 days, or scheduled for insertion within 14 days, with BIOTRONIK's most current subcutaneous cardiac rhythm monitor
* Diagnosed with paroxysmal atrial fibrillation and being evaluated for an AF ablation
* Agree to wearing a 48 hr Holter monitor
* Able and willing to complete all study visits at the study site for the study duration
* Able and willing to use a CardioMessenger® and accepts Home Monitoring concept
* Age greater than or equal to 18 years

Exclusion Criteria:

* Patient meets none of the indications for a BIOMONITOR
* Patient is planned to have an ablation prior to BIOMONITOR insertion or 48 hr Holter monitoring visit
* Patient is currently diagnosed with long-standing persistent or permanent AF
* Patient is enrolled in another study that may change or alter the cardiac rhythm that occurs prior to the completion of the Holter
* Currently indicated for or implanted with a pacemaker, ICD device, or hemodynamic monitoring system
* Life expectancy less than 6 months
* Patients reporting pregnancy at the time of enrollment

For patients enrolled after BIOMONITOR insertion:

• R-wave sensing <0.25 mV according to the most recent remote or in-person device interrogation available prior to enrollment

After the pre-Holter observation period but prior to 48 hr Holter monitoring initiation, confirm the absence of the following exclusion criteria based on the remote interrogation collected at the end of the observation period:

* No AF episodes observed or transmitted during pre-Holter observation period
* R-wave sensing <0.25 mV during pre-Holter observation period as reported by the 24 hr mean or mean value since last follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator is responsible for screening all potential subjects and selecting those who are appropriate for study inclusion. Potential subjects will be evaluated to determine if they meet the inclusion and exclusion criteria. The subjects selected for participation should be from the investigator's general patient population according to the inclusion and exclusion criteria. Patients who require a legally authorized representative will not be allowed in the study.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cardiovascular Associates, Inc., Kissimmee, Florida
  - Florida Cardiology, Winter Park, Florida
  - St. Louis Heart and Vascular, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - ProMedica Physicians Cardiology, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications, after deidentification, may be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning no later than 12 months and ending no earlier than 3 years following publication.
Access Criteria: Researchers who propose a methodologically sound proposal for analysis that is not pre-planned or already approved with another researcher and achieves aims in approved proposal, including but not limited sub-analysis or meta-analysis, will be considered. Proposals should be directed to BIOTRONIK Clinical Studies (BIOTRONIK Inc., Attn: Clinical Studies, 6024 Jean Road, Lake Oswego, OR; 1-800-547-0394). To gain access, data requestors will need to sign a data use/access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- BIOMONITOR III: Participants consented and inserted with a BIOMONITOR III
Period: Overall Study
Arm/Group | BIOMONITOR III
Started | 84
Completed | 15
Not Completed | 69
Not completed — No AF episodes detected during Pre-Holter Observation period | 49
Not completed — Study closure | 13
Not completed — Physician Decision | 3
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Mean R-wave sensing is < 0.25 mV during Pre-Holter observation period | 1

BASELINE CHARACTERISTICS:
Population: Baseline data collected from all participants consented and inserted with a BIOMONITOR III, when available.
Arm/Group | BIOMONITOR III
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 64
  More than one race | 0
  Unknown or Not Reported | 8
Height [Mean (Standard Deviation); unit: Inches] | 67.8 (4.8)
Weight [Mean (Standard Deviation); unit: Pounds] | 220.9 (53.0)

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Sensitivity
Description: The diagnostic sensitivity of the BIOMONITOR will be determined by comparing AF events detected by the BIOMONITOR and 48 hr Holter monitor for each subject. Diagnostic sensitivity is the ability of the BIOMONITOR to correctly identify subjects who have true AF as determined by the Holter monitor. It is calculated as the number of participants with a true BIOMONITOR AF detection divided by the sum of the number of participants with a true BIOMONITOR AF detection and the number of participants with a false negative BIOMONITOR AF detection.
Time Frame: 48 hours
Population: Participants with an evaluable Holter recording who have completed the 48 hr Holter monitor
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOMONITOR III
Number analyzed (Participants) | 25
percentage of participants | 90.9 [71 to 100]

ADVERSE EVENTS:
Time Frame: Insertion through study exit or study termination, an average of 1.7 months, and up to 5.7 months
Description: Sites were required to report all insertion procedure-related and device-related adverse events. Additionally, sites were required to report all non-procedure non-system related adverse events if any of the following occur and require device removal: (1) Secondary infection, and (2) Other non-elective intervention
Arm/Group | BIOMONITOR III
All-Cause Mortality (participants affected / at risk) | 1/84
Serious Adverse Events (participants affected / at risk) | 1/84
Other Adverse Events (participants affected / at risk) | 1/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOMONITOR III (N=84)
Surgical site infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOMONITOR III (N=84)
Cellulitis at implant site (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT04076917/Prot_000.pdf